CLINICAL TRIAL: NCT02516839
Title: Treatment of Obesity Targeting Appetite and Cue Reactivity
Brief Title: PACIFIC: Providing Adults Collaborative Interventions For Ideal Changes
Acronym: ROC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151110; 1R01DK103554-01A1 (NIH)
Record Dates: First submitted 2015-07-31; First posted 2015-08-06 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Overeating; Body Mass Index; Weight; Treatment; Cravings; Intervention; Behavioral Treatment
MeSH Terms: conditions — Overweight; Obesity; Hyperphagia; Body Weight | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regulation of Cues (ROC) (Experimental): The ROC program provides psychoeducation, coping skills, self-monitoring and experiential learning.
  Interventions: Behavioral: Regulation of Cues (ROC)
- Behavioral Weight Loss (BWL) (Experimental): The BWL program will include dietary recommendations, physical activity recommendations, and behavioral change recommendations.
  Interventions: Behavioral: Behavioral Weight Loss (BWL)
- BWL+ ROC (Experimental): BWL and ROC will be integrated for this arm, to capitalize on the strengths of both treatments.
  Interventions: Behavioral: BWL + ROC
- Nutrition Education, Stress Management Social Support (Active Comparator): Nutrition Education, Stress Management and Social Support will be covered. Mindfulness will be practiced in every session.
  Interventions: Behavioral: Nutrition Education, Stress Management and Social Support

INTERVENTIONS:
Behavioral: Regulation of Cues (ROC) — Participants are provided information about basic learning theory and how physiological responses to food cues develop and can be managed. Lack of sensitivity to appetite and satiety cues and increased sensitivity to food cues will be discussed. Coping skills are presented to assist in mastery and toleration of food cue sensitivity. Participants will complete experiential learning exercises with food, and taught to monitor their hunger,satiety, and cravings. The physical activity program will focus on increasing both lifestyle activity and structured exercise programs.
  Other Names: ROC
  Arms: Regulation of Cues (ROC)
Behavioral: Behavioral Weight Loss (BWL) — All participants will be instructed on how to consume a balanced deficit diet of conventional foods; individual goals for energy intake will be based on initial body weight. Participants will be instructed in measuring portion sizes, counting calories (with a calorie counter provided or on their phone), and self-monitoring food intake. The physical activity program will focus on increasing both lifestyle activity and structured exercise programs. Behavior change recommendations include stimulus control, self-monitoring, goal setting, managing high-risk situations, meal planning, slowing eating, problem solving, social support, cognitive restructuring, lapse and relapse prevention skills, and maintaining weight loss.
  Other Names: BWL
  Arms: Behavioral Weight Loss (BWL)
Behavioral: BWL + ROC — BWL and ROC will be integrated for this arm, to capitalize on the strengths of both treatments. All participants will be taught to decrease caloric intake and increase physical activity, and to use all of the behavioral skills provided in BWL. However, they will also be taught models of hunger and satiety and about food cue reactivity, and will learn skills to manage these. This arm will include an experiential component, including hunger monitoring during dinner and participating in exposure sessions in the clinic.
  Arms: BWL+ ROC
Behavioral: Nutrition Education, Stress Management and Social Support — Topics included will be stress management/relaxation, social support, and nutrition education. There will be a strong mindfulness component to this group.
  Arms: Nutrition Education, Stress Management Social Support

SUMMARY:
The objective of this proposed study is to collect initial efficacy data on ROC and ROC + BWL compared to an active comparator (AC) and to BWL.

DETAILED DESCRIPTION:
The investigators have developed a new model for the treatment of obesity, called Regulation of Cues (ROC), which is based on Schachter's Externality Theory. The ROC program targets two theorized mechanisms for overeating in Schachter's Theory; decreased sensitivity to appetitive cues and increased sensitivity to external food cues. Considering that BWL has merit for some people, but fails to facilitate maintenance, this study will compare ROC, BWL, ROC+BWL combined and an active comparator (AC). The investigators will recruit overweight/obese adults and will assess them at baseline, mid-treatment (month 6), post-treatment (month 12), mid-follow-up (month 18) and follow-up (month 24). Assessments will include body mass index (BMI), body composition, and binge eating over the course of treatment and follow-up. This study will contribute to the study of basic behavioral mechanisms and food intake, could provide a novel model for the treatment of obesity, and could inform clinical decision making regarding obesity treatment.

ELIGIBILITY:
1. All participants will be between the ages of 18-65 meeting criteria for overweight, with a BMI between 25 and 45.
2. Participants will provide written informed consent for study participation.
3. Participants will possess English language skills at the 5th grade reading level.
4. Participants will be free of major medical conditions such as a recent history of coronary heart disease; recent history of myocardial infarction; recent symptoms of angina, diabetes, recent stroke, orthopedic problems that would limit activity during the following twelve months; or any other serious medical condition that would make physical activity unsafe.
5. Participants will not have bulimia or anorexia, significant cognitive impairment, a known psychotic disorder, or unstable psychiatric illness (e.g., recent psychiatric hospitalization, acute suicidal ideation) as derived from their intake interview and questionnaires.
6. Participants will not be moving out of the San Diego area for the duration of their study enrollment (24 months).
7. Participants will not be pregnant, planning to get pregnant in the 2 year study period or lactating.
8. Participants will not be taking medication for weight loss or that may impair physical activity tolerance or performance.
9. Participants with medical or psychological problems, or taking medications that could make adherence with the study protocol difficult or dangerous will not be included.
10. Participants cannot have a history of bariatric surgery
11. Participants cannot currently be enrolled in an organized weight control program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2015-09; Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
body mass index as measured by height and weight | Time Frame: Change from baseline at an average of 12 months and 24 months
binge eating as measured by the Eating Disorder Examination | Change from baseline at an average of 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — UCSD
Locations (1):
- UCSD Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California, United States

REFERENCES:
- [Background] Boutelle KN, Zucker NL, Peterson CB, Rydell SA, Cafri G, Harnack L. Two novel treatments to reduce overeating in overweight children: a randomized controlled trial. J Consult Clin Psychol. 2011 Dec;79(6):759-71. doi: 10.1037/a0025713. PMID 22122291
- [Background] Boutelle KN, Zucker N, Peterson CB, Rydell S, Carlson J, Harnack LJ. An intervention based on Schachter's externality theory for overweight children: the regulation of cues pilot. J Pediatr Psychol. 2014 May;39(4):405-17. doi: 10.1093/jpepsy/jst142. Epub 2014 Jan 23. PMID 24459240
- [Derived] Boutelle KN, Pasquale EK, Strong DR, Eichen DM, Peterson CB. Reduction in eating disorder symptoms among adults in different weight loss interventions. Eat Behav. 2023 Dec;51:101787. doi: 10.1016/j.eatbeh.2023.101787. Epub 2023 Jul 24. PMID 37639734
- [Derived] Boutelle KN, Eichen DM, Peterson CB, Strong DR, Kang-Sim DE, Rock CL, Marcus BH. Effect of a Novel Intervention Targeting Appetitive Traits on Body Mass Index Among Adults With Overweight or Obesity: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2212354. doi: 10.1001/jamanetworkopen.2022.12354. PMID 35583870